CLINICAL TRIAL: NCT00109434
Title: The Effect of Exercise on the Development of Hypoglycemia in Children With Type 1 Diabetes; A Study Being Conducted by the Diabetes Research in Children Network
Brief Title: Study to Determine the Relationship Between Exercise and Hypoglycemia in Children With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: DirecNet 005; HD41890
Record Dates: First submitted 2005-04-27; First posted 2005-04-28 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Type I
Keywords: exercise; hypoglycemia; Diabetes Mellitus, Type I; glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The main purpose of this study is to find out how often low blood sugar (hypoglycemia) happens during the night after exercise in the late afternoon. The study also will see if there are any factors that can predict if low blood sugar is going to develop. Blood samples will also be drawn to measure two hormones-glucagon and epinephrine (adrenaline)-to see how they are affected by exercise. Glucagon helps to raise the blood sugar when it is low. Epinephrine causes symptoms that make the person aware that the blood sugar is low. From the blood sample, other substances in the blood may also be measured to see how they are affected by exercise.

A second purpose of the study is to find out whether exercise affects the accuracy of a continuous glucose sensor (CGMS made by Medtronic Minimed).

The study will also look at the accuracy of different home glucose meters.

DETAILED DESCRIPTION:
Many children and adults with type 1 diabetes have a drop in the blood sugar during exercise. When someone has low blood sugar, the body tries to return the blood sugar to normal. Some studies show that after exercise, the blood sugar may drop later in the day or during the night. However, it is not known how often this happens. Also, not enough is known about how exercise affects blood sugar or the awareness of low blood sugar.

Some studies in adults have shown that exercise may affect the body's natural response to low blood sugar and exercise in the future.

For this study, each subject will have two in-patient hospital stays 1 to 4 weeks apart, each lasting about 24 hours: one with no exercise and one with a 75-minute exercise session in the late afternoon. (The order of the exercise and sedentary days will be determined at random.)

Prior to each hospital admission, each subject will keep a detailed diary of insulin use and hypoglycemia for one week.

On each of the two admissions, the insulin regimens and diet will be as similar as possible.

On each of the 2 admissions, the following will occur:

* A CGMS sensor will be inserted and calibrated.
* An intravenous catheter for the collection of blood samples will be inserted.
* Blood sugar measurements will be made with an Ultra, BD Logic, and Freestyle meter every half hour beginning at 10:00 p.m. through 6:00 a.m.
* Blood samples for glucagon, epinephrine, and glucose will be collected hourly from 10:00 p.m. to 6:00 a.m.

On the exercise day only,

* In the morning, the subject will run on the treadmill for about 5 minutes to determine the settings needed to achieve a heart rate of 140.
* Exercise will begin at approximately 4:00PM and will consist of 15 minutes on a treadmill at a heart rate of approximately 140 followed by a 5-minute rest period. This cycle will be repeated 3 more times for a total of four 15-minute exercise periods with 5-minute rest periods in between (75 minutes total). A heart rate monitor will be worn throughout the time of exercise to ascertain the effort put forth.
* BG (blood glucose) measurements will be made using the Ultra, BD Logic, and Freestyle meters (1) prior to starting the exercise, (2) during each of the 3 rest periods, (3) immediately following the exercise session, and (4) at 15 minute intervals for one hour following the completion of the exercise. Blood samples will be collected for the central lab at the times of sampling for glucagon and epinephrine.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes for at least 18 months
* HbA1c <10.0% as measured by the DCA2000.
* Age 10.0 to <18.0 years
* Weight >36.0 kg
* BMI (body mass index) >5th and <95th percentiles for age/gender
* Stable insulin regimen for at least 1 month and not anticipating a change prior to the subject's completion of the study
* Insulin regimen involves either use of an insulin pump or Lantus (with short-acting insulin)
* NPH or Lente, if part of the insulin regimen, is given only in the morning before breakfast
* Normal hematocrit (within normal limits of local laboratory)
* Normal thyroid function (measured within the previous year)
* Parent/guardian and subject understand the study protocol and agree to comply with it
* Informed Consent Form signed by the parent/guardian and Child Assent Form signed

Exclusion Criteria:

* Insulin regimen includes Ultralente/Lente or NPH at times other than the morning before breakfast
* A recent injury to body or limb, Addison's disease, muscular disorder, use of any medication or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the exercise protocol
* Asthma which has been medically treated within the last year
* Current use of glucocorticoid medication (by any route of administration)
* Current use of a beta blocker medication
* Use of pseudoephedrine 48 hours prior to CRC admission (if used in the 48 hours prior to the scheduled second admission, the admission will be deferred)
* Severe hypoglycemia resulting in seizure or loss of consciousness in the 2 weeks prior to CRC admission (if a severe episode occurs within 2 weeks prior to the scheduled second admission, the admission will be deferred)
* Active infection (if at the time of the planned second admission an infection is present, the admission will be deferred)
* Anticipating a significant change in exercise regimen between admissions (i.e. starting or stopping an organized sport)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Start 2004-06; Study Completion 2004-11

PRIMARY OUTCOMES:
Hypoglycemia defined as <=70 mg/dL.

SECONDARY OUTCOMES:
Changes in epinephrine and glucagon levels.

CONTACTS AND LOCATIONS:
Overall Officials: William V Tamborlane, M.D., Study Chair — Department of Pediatrics, Yale University School of Medicine
Locations (5):
- United States (5):
  - Division of Pediatric Endocrinology and Diabetes, Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, University of Colorado, Denver, Colorado
  - Department of Pediatrics, Yale University School of Medicine, New Haven, Connecticut
  - Nemours Children's Clinic, Jacksonville, Florida
  - Department of Pediatrics, University of Iowa Carver College of Medicine, Iowa City, Iowa

REFERENCES:
- [Background] Tsalikian E, Mauras N, Beck RW, Tamborlane WV, Janz KF, Chase HP, Wysocki T, Weinzimer SA, Buckingham BA, Kollman C, Xing D, Ruedy KJ; Diabetes Research In Children Network Direcnet Study Group. Impact of exercise on overnight glycemic control in children with type 1 diabetes mellitus. J Pediatr. 2005 Oct;147(4):528-34. doi: 10.1016/j.jpeds.2005.04.065. PMID 16227041
- [Result] Weinzimer SA, Beck RW, Chase HP, Fox LA, Buckingham BA, Tamborlane WV, Kollman C, Coffey J, Xing D, Ruedy KJ; Diabetes Research in Children Network Study Group. Accuracy of newer-generation home blood glucose meters in a Diabetes Research in Children Network (DirecNet) inpatient exercise study. Diabetes Technol Ther. 2005 Oct;7(5):675-80; discussion 681-3. doi: 10.1089/dia.2005.7.675. PMID 16241867
- [Result] Diabetes Research in Children Network (DirecNet) Study Group. Impaired overnight counterregulatory hormone responses to spontaneous hypoglycemia in children with type 1 diabetes. Pediatr Diabetes. 2007 Aug;8(4):199-205. doi: 10.1111/j.1399-5448.2007.00248.x. PMID 17659061
- [Result] Diabetes Research In Children Network (Direcnet) Study Group; Buckingham BA, Kollman C, Beck R, Kalajian A, Fiallo-Scharer R, Tansey MJ, Fox LA, Wilson DM, Weinzimer SA, Ruedy KJ, Tamborlane WV. Evaluation of factors affecting CGMS calibration. Diabetes Technol Ther. 2006 Jun;8(3):318-25. doi: 10.1089/dia.2006.8.318. PMID 16800753
- [Result] Tansey MJ, Tsalikian E, Beck RW, Mauras N, Buckingham BA, Weinzimer SA, Janz KF, Kollman C, Xing D, Ruedy KJ, Steffes MW, Borland TM, Singh RJ, Tamborlane WV; Diabetes Research in Children Network (DirecNet) Study Group. The effects of aerobic exercise on glucose and counterregulatory hormone concentrations in children with type 1 diabetes. Diabetes Care. 2006 Jan;29(1):20-5. doi: 10.2337/diacare.29.1.20. PMID 16373890